CLINICAL TRIAL: NCT01683292
Title: An Ascending-Dose, Single-Centre Study Investigating the Safety, Tolerability, Efficacy, and Pharmacokinetics of VR040(Inhaled Apomorphine)in Parkinson's Disease
Brief Title: Single-Centre Study of VR040(Inhaled Apomorphine) in Idiopathic Parkinson's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: South Glasgow University Hospitals NHS Trust (Other)
Collaborators: Vectura Limited (Industry)
Responsible Party: Principal Investigator, Dr Donald Grosset, Consultant Neurologist, South Glasgow University Hospitals NHS Trust
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VR040/001
Record Dates: First submitted 2012-09-07; First posted 2012-09-11 (Estimated); Last update posted 2012-09-11 (Estimated); Status verified 2012-09

CONDITIONS: Parkinson's Disease
Keywords: apomorphine; inhaled; motor fluctuations
MeSH Terms: conditions — Parkinson Disease; Respiratory Aspiration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Inhaled VR040 (Experimental): Inhaled apomorphine, dry powder, VR040 at fine particle doses (FPD) of 0.2mg, 0.5mg and 0.8mg. A single dose, followed by a second dose at 12 minutes if efficacy end point was not attained.
  Interventions: Drug: Inhaled VR040
- Placebo (Placebo Comparator): Inhaled dry powder. A single dose, followed by a second dose at 12 minutes if efficacy end point was not attained.
  Interventions: Drug: Placebo for VR040

INTERVENTIONS:
Drug: Inhaled VR040
  Other Names: Inhaled apomorphine
  Arms: Inhaled VR040
Drug: Placebo for VR040 — Placebo arm
  Arms: Placebo

SUMMARY:
In this first study of inhaled apomorphine in Parkinson's disease patients, the primary objective is to find the minimum efficacious dose of apomorphine that is useful in rescuing patients during 'off' periods. Safety, tolerability and pharmacokinetics of inhaled apomorphine will be assessed during the study.

DETAILED DESCRIPTION:
Objectives:

ELIGIBILITY:
Inclusion Criteria:

1. Patients with established idiopathic PD (via fulfilment of Steps 1 and 2 of the UK Brain Bank Criteria), of at least 3 years duration prior to study entry, who were on specific and optimised anti-Parkinson medication (levodopa and/or dopamine agonists), and with motor fluctuations.
2. Patients with a modified Hoehn and Yahr disease severity scoring of between 2 and 4 in an "on" state.
3. Men or women aged over 30 years.
4. Patients with a signed and dated written valid consent obtained prior to participation.
5. Female patients must have been of non-childbearing potential (ie, physiologically incapable of becoming pregnant, including any female who was post-menopausal) or of child-bearing potential with a negative pregnancy test (urine or serum) at screening.
6. Patients who experienced motor fluctuations with recognisable "off" periods in control of motor symptoms, as assessed by the motor fluctuation questionnaire (patients were to have reported at least 1 "Yes" response to the questions in the motor fluctuation questionnaire).
7. Patient willing and able to comply with study procedures.-

Exclusion Criteria:

1. Patients who had participated in a trial with an investigational product within 3 months prior to randomisation at Visit 2.
2. Patients with serious uncontrolled disease including serious psychological disorders likely to interfere with the study and/or likely to cause death within 6 months of the study completion.
3. Patients with previous intolerance to apomorphine.
4. Patients with a previous significant complication from oral dopamine agonist therapy including hospitalisation following dopamine agonist introduction and/or the development of hallucinations or other adverse neuropsychiatric features following introduction of sc apomorphine.
5. Women lactating, pregnant, or of child-bearing potential not using a reliable contraceptive method.
6. Patients with known HIV or active chronic hepatitis B or C infection.
7. Patients with any clinically significant abnormality following review of screening laboratory data and full physical examination.
8. Patients who, in the Investigator's opinion, were unsuitable for the study for any reason.
9. Patients with clinically significant blood test abnormalities and previous medical history/intercurrent illnesses that may have compromised the safety of the patient in the study.
10. Patients with major ECG abnormalities (as judged by the Investigator).
11. Patients with a FEV1 <65%.
12. Patients showing a postural decrease in systolic blood pressure (BP) of > 20 mm Hg, or showing significant clinical symptoms associated with orthostatic hypotension.
13. Patients with persistent elevation of BP, with average systolic readings of 160 mm Hg or average diastolic readings of 100 mm Hg.
14. Patients taking anabolic steroids, traditional antipsychotics (unless low dose), and antiemetics other than domperidone.
15. Patients taking agents of the 5HT3 antagonist class including ondansetron, granisetron, dolasetron, palonosetron, and alosetron.
16. Patients with existing cancer and those in remission for less than 5 years.
17. Patients with evidence (as ascertained from examination, tests or history) to indicate cardiovascular, gastrointestinal tract, liver, kidney, central nervous system, pulmonary system, or bone marrow disorders that in the Investigator's opinion compromised patient safety.
18. Patients who were known non-responders to apomorphine treatment for "off" episodes.
19. Patients with a history of drug or alcohol abuse in the 12 months prior to entry.
20. Patients with a history of clinically significant allergies to VR040 formulation constituents (including lactose and opioids) and domperidone.
21. Patients with signs or symptoms suggestive of schizophrenia, dementia, "Parkinson plus" syndromes, or unstable systemic disease

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2006-01; Primary Completion 2006-06 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
The proportion of patients "on" at any time post-dosing. | up to 80 minutes
  Parkinson's motor severity assessed by a clinician, and disease state assessment by the patient, were performed at baseline during an 'off' state, and at specified times after test drug administration.

SECONDARY OUTCOMES:
Duration that patients remain in an "on" state. | until return to "off" up to 3 hours
  Time from when patient switched "on" after inhalation of study product, until patient returned to "off" state.

CONTACTS AND LOCATIONS:
Locations (1):
- Southern General Hospital, Glasgow, United Kingdom